CLINICAL TRIAL: NCT03593512
Title: Deep Brain Stimulation for Autonomic and Gait Symptoms in Multiple System Atrophy
Acronym: STAG-MSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13340
Record Dates: First submitted 2018-05-22; First posted 2018-07-20 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-05

CONDITIONS: Multiple System Atrophy; Autonomic Failure; Postural Hypotension; Bladder, Neurogenic; Gait Disorders, Neurologic
Keywords: multiple system atrophy; autonomic
MeSH Terms: conditions — Multiple System Atrophy; Pure Autonomic Failure; Hypotension, Orthostatic; Urinary Bladder, Neurogenic; Gait Disorders, Neurologic | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Evaluation of symptomatology before and after implantation of DBS electrodes; followed by cross-over of "on" and "off" stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PPN DBS (Experimental): All patients will undergo bilateral PPN DBS
  Interventions: Procedure: Deep brain stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation — Bilateral deep brain stimulation of the pedunculopontine nucleus

SUMMARY:
Patients referred to neurosurgery routinely and safely undergo deep brain stimulation (DBS) for treatment of symptoms related to neurodegenerative conditions, most commonly Parkinson's disease.

In the investigators experience, and published evidence shows, that stimulation has effects on the autonomic nervous system. In patients undergoing therapeutic DBS for a particular subtype of Parkinsonism, Multiple System Atrophy, the further effects on autonomic parameters such as blood pressure and bladder symptoms as well as the originally intended indications (gait and movement disorder) will be investigated. The mechanisms of any effects will also be studied by using a number of techniques such as magnetoencephalography (MEG) and Muscle Sympathetic Nerve Activity (MSNA) recording.

Key goals are to:

1. Demonstrate that stimulation of the peduculopontine nucleus (PPN) improves autonomic function and has an attendant improvement on patients' quality of life
2. Investigate the role of the PPN and how it interacts with other brain areas.

This translational strategy will lead to a larger efficacy study of DBS for MSA as well as revolutionizing neural-based treatments in other autonomic disorders such as orthostatic hypotension and pure autonomic failure.

DETAILED DESCRIPTION:
AIMS OF THE PROJECT AND IMPORTANCE

Multiple system atrophy (MSA) is a form of Parkinsonism and is a neurodegenerative condition that is characterized by gait and autonomic failure. MSA symptoms are generally poorly responsive to medicines that treat Parkinson's disease (PD), and so symptom control is difficult.

The aim is to assess the effects of deep brain stimulation (DBS) of the pedunculopontine nucleus (PPN) on autonomic and gait symptoms to show that it improves quality of life in patients with MSA.

Secondary aims are to assess the effects of stimulation on autonomic parameters (cardiovascular and bladder function) as well as the routine parameters of the movement disorder (gait, freezing and falls, etc).

In addition, there is a mechanistic component of the study looking at both peripheral autonomic activity and brain networks associated with stimulation.

BACKGROUND AND WORK LEADING UP TO THE PROJECT

DBS is a routine treatment for movement disorders such as Parkinson's disease and dystonia. MSA is a 'Parkinsonian' condition similar to PD and is a progressive, incurable, neurodegenerative condition characterized by a combination of Parkinsonism, ataxia, and autonomic failure. Autonomic dysfunction is the presenting feature in half of patients that have Parkinsonism or ataxia predominant MSA.

Whilst DBS is sometimes performed for the treatment of MSA, the primary outcome measure is usually the motor outcome, despite the fact that the autonomic symptoms may be the predominant factor in causing a reduced quality of life. This is because DBS is traditionally used to control motor symptoms and the exploration of its effects on autonomic function are relatively new, and pioneered by our group. The most common complaints caused by autonomic dysfunction in MSA are related to orthostatic hypotension and neurogenic bladder, both of which have been studied by the investigators previously.

Part of the aim of this study is to look at orthostatic BP changes with and without stimulation and see whether these are improved by DBS. Bladder dysfunction includes incontinence and incomplete emptying. These will be investigated using urodynamic testing, with a standard protocol. Other 'autonomic' problems include sleep disorders, exercise intolerance and problems with thermoregulation and sweating. These will be captured using questionnaires.

Regarding the target used for DBS, a well-established target to improve gait and postural abnormalities in PD is the pedunculopontine nucleus (PPN). The investigators have previously demonstrated that the PPN is also a brain area that, when stimulated, improves bladder function in these patients. They have also shown (unpublished data) that PPN stimulation reduces postural fall in BP in a group of PD patients treated primarily for gait and postural problems. It has also been shown that stimulation of a related brain area can improve orthostatic hypotension.

Mechanistic Studies

These are important in order to understand how PPN DBS alters autonomic function. Previously, the investigators have studied the effects of central stimulation of the subthalamic nucleus and periaqueductal grey area (amongst others) on peripheral sympathetic nerve activity. These techniques (muscle sympathetic nerve activity (MSNA)) will be applied in the current study to find out whether PPN DBS alters peripheral sympathetic nervous system activity.

To look at central mechanisms, two techniques will be used. Firstly, diffusion tensor imaging is routinely obtained as part of surgical planning. The hypothesis is that connections from PPN to areas that are part of the central autonomic network are important for influencing autonomic control. By looking at tracts to and from the target area, it will be investigated whether connections to the rostroventrolateral medulla (RVLM) are important for changes in MSNA. The RVLM is an important area that receives feedback from the periphery and is in turn influenced by higher centres.

A second part of the central mechanism study will utilize MEG scanning. The investigators have previously applied this technique to patients who have undergone DBS. The investigator are interested in whether PPN DBS alters cortical activity, both in the insula and anterior cingulate cortices (these are important in autonomic control) and also the motor cortex (important for motor control).

KEY METHODOLOGIES AND TECHNIQUES

Recruitment

Patients will be identified in a movement disorder clinic by a consultant neurologist. If they decide to take part, they will attend to proceed with the consent process and baseline measurements. The pathway for each participant through the study will follow a standardized pattern that is essentially identical to the pathway that current DBS patients for all movement disorder indications go through.

Baseline Assessments

1. Questionnaires

   1. EQ-5D - quality of life questionnaire
   2. UMSARS - Unified MSA rating scale
   3. Freezing of Gait (FOG) Questionnaire
   4. Autonomic questionnaire
   5. Falls diary
2. Neuropsychology assessment. Includes HAD, FLP and MOCA questionnaires and interview.
3. MRI scan with DTI. This is routine for surgical planning.
4. Gait analysis. Patients will be asked to walk along a special gait flooring which will allow us to obtain specific parameters concerning their gait.
5. Urodynamics and Cardiovascular tests

   1. Urodynamics

      The 'gold standard' is video urodynamics. This involves urethral catheterisation and insertion of a rectal probe and measurements of detrusor pressures, bladder capacity, reflux, sensory urgency and voiding differences such as rate of urinary flow. Patients who are unwilling to undergo these tests will still fill in voiding diaries and urinary symptom questionnaires that are part of the questionnaires listed above.
   2. Tilt table tests

      Patients will undergo continuous ECG monitoring whilst standing upright and then whilst tilted into a lying down position using the tilt table. Changes in heart rate, heart rate variability and blood pressure will be recorded and integrated using our analysis program.
   3. Ambulatory BP

This involves wearing a blood pressure cuff for 24 hours, which will be timed with the other baseline assessments or, if the participant prefers, this can be done at home.

Subsequent Visits

1. Surgery

   This will follow routine clinical practice. Electrodes will be implanted under general anaesthetic using a standard stereotactic frame. Electrodes will be externalized for a week of clinical testing. During the week of testing, the priority will be to titrate the stimulator for clinical effects. Further gait analysis, tilt table tests and ambulatory BP may be used to inform parameter settings. In addition, we may perform local field potential recordings (recording electrical activity from the electrodes) during these tests. This will give information as to how the PPN is responding to movement and tilt etc. At the end of one week, a second procedure will be performed to insert the implantable pulse generator (the battery). They will return at 6 weeks for stimulator titration only (this is part of routine care).
2. 3 month primary outcome follow up

   1. Questionnaires (section 1 and 2 in baseline assessments above) will be performed as at baseline except the full neuropsychology assessment will not be performed (just the HADS, FLP and MOCA).
   2. The following tests will be repeated on and off stimulation; i) Urodynamics ii) Tilt table tests iii) Gait analysis
   3. The participants will attend for a second day and will undergo two further tests ON and OFF stimulation

   i. Magnetoencephalography (MEG) scan. This records cortical signals ON and OFF stimulation with the aim of demonstrating how PPN suppression or excitation alters cortical activity, especially in the areas important for autonomic and motor control ii. MSNA (microneurography). This technique entails insertion of two very fine needles (30-40microns in diameter) below the knee. The first will record directly from the common peroneal nerve whilst the second will lie subcutaneously as a reference. This is an established technique for measuring peripheral sympathetic activity. Neurograms will be recorded with stimulation ON and then OFF during the same sitting. The aim is to establish whether any changes in autonomic symptomatology are correlated with changes in sympathetic nerve activity, thereby providing a mechanism of action.

   iii. Sleep EEG studies with varying stimulation ON and OFF in order to investigate the role of the PPN in sleep stages and EEG waveforms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MSA with disabling autonomic symptoms (bladder dysfunction and orthostatic symptoms
2. UMSARS score of >40
3. >6/12 in the autonomic subsection (Q9-12) of the UMSAR scale
4. Patient willing and able to give informed consent to involvement in the study.
5. Male or female, aged 18 years or over.
6. Able to walk unaided (to perform gait analysis)
7. Have an anticipated prognosis > 2 years

Exclusion Criteria:

1. The patient is unwilling to participate or unable to give informed consent.
2. The patient has been deemed unfit for stimulator insertion by their healthcare team i.e. surgical contraindications to DBS:

   * Bleeding or coagulation disorder
   * Not fit for general anaesthetic
   * Unable to deal with implanted DBS system (turn on and off and recharging where applicable, although it is acceptable if a carer can do this)
3. Untreated anxiety or depression
4. Unable to undergo MRI (eg. metal implants)
5. Subject is currently participating in a clinical investigation that includes an active treatment arm.
6. Female who is pregnant - testing will be offered to female patients who are unsure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
EuroQol 5 Dimension (5 level) score before and after deep brain stimulation | Through study completion, but on average, over an 8 month period for each patient
  Measurement of quality of life before and after surgery. Results will be given as description of health states - it is not quantitative.
Fluency of gait as measured by accelerometry before and after deep brain stimulation | Through study completion, but on average, over an 8 month period for each patient
  Measurement of gait parameters before and after surgery
Modified composite autonomic symptom scale before and after deep brains stimulation | Through study completion, but on average, over an 8 month period for each patient
  Measurement of autonomic symptomatology before and after surgery - Score from 0-100
Change in postural blood pressure change before and after PPN DBS | Through study completion, but on average, over an 8 month period for each patient
  Measurement of effect on postural blood pressure change before and after surgery

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by using approved UK reporting procedure | Through study completion, 2 years
  To assess the safety of PPN DBS on MSA patients by recording adverse events
Muscle sympathetic nerve activity before and after deep brain stimulation | Through study completion, but on average, over an 8 month period for each patient
  To determine whether or not PPN suppression or excitation alters sympathetic outflow by measuring the activity in autonomic nerves in the leg
Cortical magentoencephalography profile with deep brain stimulation on and off | 3-6 months after surgery
  Identification in change of cortical magetic activity with DBS on and off
Physical anatomical white matter connections between the pedunculopontine nucleus and the rest of the central nervous system | Before surgery and 3-6 months after surgery
  To identify the physical anatomical relations of the stimulated region of brain by looking at high resolution structural imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Alex L Green, FRCS(SN), Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We are recruiting only 10 patients, so sharing IPD even anonymised, may be identifiable. Decision will be taken when this can be definitively elucidated.